CLINICAL TRIAL: NCT02450643
Title: Evaluation of Hypoallergenicity of a New Extensively Hydrolyzed Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 14.24.CLI
Record Dates: First submitted 2015-05-07; First posted 2015-05-21 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Cow's Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test then Control (Active Comparator): Subjects will perform a DBPCFC with the Test formula followed by the Control formula
  Interventions: Other: Test extensively hydrolyzed formula; Other: Control extensively hydrolyzed formula
- Control then Test (Active Comparator): Subjects will perform a DBPCFC with the Control formula followed by the Test formula
  Interventions: Other: Test extensively hydrolyzed formula; Other: Control extensively hydrolyzed formula

INTERVENTIONS:
Other: Test extensively hydrolyzed formula — extensively hydrolyzed formula made with a new enzyme
Other: Control extensively hydrolyzed formula — commercially available extensively hydrolyzed formula

SUMMARY:
Infants/children with cow's milk allergy will take part in 2 double-blinded placebo-controlled food challenges (DBPCFC) of 2 extensively hydrolyzed formulas in random order. If both food challenges are passed, subjects will be asked to consume the Test formula in an at-home open challenge for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Born at term (>36 weeks gestation)
* 2 months to <4 years of age at enrollment
* Documented CMA within 6 months prior to enrollment
* Otherwise healthy
* Having obtained his/her legal representative's informed consent

Exclusion Criteria:

* Children consuming mother's milk at the time of inclusion and during the trial
* Any chromosomal or major congenital anomalies
* Chronic medical diseases (ie seizure disorders, chronic lung disease, heart problems (heart murmurs okay))
* Immunodeficiency
* Receiving free amino acid formula
* Subject who in the Investigator's assessment cannot be expected to adhere to the study protocol
* Currently participating in another clinical trial.

Ages: 2 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 83 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
allergic reaction | 2 hours post-DBPCFC
  number of children who react during a DBPCFC to either formula

SECONDARY OUTCOMES:
stool characteristics | 1 week
  stool descriptors as collected on daily diaries
formula intake | 1 week
  amount of formula ingested as collected on daily diaries
adverse events | 1 week
  any adverse event reported by caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nowak-Wegrzyn, MD, Principal Investigator — Mt. Sinai
Locations (8):
- United States (8):
  - Atria Clinical Research, Little Rock, Arkansas
  - Allergy and Asthma Associates of Southern California, Mission Viejo, California
  - All Children's Hospital, St. Petersburg, Florida
  - AeroAllergy, Savannah, Georgia
  - Mt. Sinai, New York, New York
  - ENT & Allergy Associates, Newburgh, New York
  - Allergy and Sinus Relief Center/Great Lakes Medical research, Chardon, Ohio
  - Allergy Asthma Research Institute, Waco, Texas